CLINICAL TRIAL: NCT06972186
Title: Neuromotor Adaptation to Fatigue: Changes in Lower Extremity Proprioception in Patients With Osteoarthritis
Brief Title: Proprioceptive Fatigue Adaptation in Osteoarthritis
Acronym: PROFA-OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KOSTU-25-OA-01
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis of Knee; Proprioception; Isokinetic Test; Gonarthritis
Keywords: osteoarthritis of knee; propripception; isokinetic test; gonarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Active Comparator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Control (Active Comparator): Age- and sex-matched postmenopausal women without knee pathology. Participants will perform the same passive and active joint position sense tests as the gonarthrosis group, before and after a control fatigue protocol using the Biodex system.
  Interventions: Diagnostic Test: Fatigue Protocol + Joint Position Sense Testing
- Gonarthrosis Group (Experimental): Postmenopausal women aged 50-65 with Kellgren-Lawrence Grade 2-3 knee osteoarthritis.
  Participants will undergo an isokinetic fatigue protocol at 180°/s using a Biodex dynamometer. Passive and active joint position sense tests will be performed before and after fatigue.
  Interventions: Diagnostic Test: Fatigue Protocol + Joint Position Sense Testing

INTERVENTIONS:
Diagnostic Test: Fatigue Protocol + Joint Position Sense Testing — Groups will undergo an isokinetic fatigue protocol at 180°/s using a Biodex dynamometer. Passive and active joint position sense tests will be performed before and after fatigue.

SUMMARY:
This study aims to investigate the effects of fatigue induced by isokinetic exercise on passive and active joint position sense in postmenopausal women diagnosed with knee osteoarthritis (gonarthrosis). A healthy control group matched for age and sex will also be included for comparative analysis. Participants will undergo proprioceptive assessments before and after an isokinetic fatigue protocol. We hypothesize that (1) fatigue will impair both passive and active joint position sense in patients with gonarthrosis, (2) active joint position sense will be more affected than passive sense, and (3) the deterioration in proprioception will be greater in the gonarthrosis group compared to healthy controls.

DETAILED DESCRIPTION:
Osteoarthritis, particularly knee osteoarthritis (gonarthrosis), is a progressive musculoskeletal disease that severely affects lower extremity functions. Proprioceptive impairments in these patients can lead to altered motor control, reduced movement accuracy, and increased risk of falls. Fatigue may exacerbate these impairments by affecting sensory feedback from muscle spindles and joint receptors, which is critical for joint stability and motor control. In postmenopausal women, hormonal changes further compound muscle weakness and joint instability, highlighting the clinical importance of understanding proprioceptive changes following fatigue.

This experimental study will involve two groups: postmenopausal women with gonarthrosis and age-matched healthy controls. Participants will undergo an isokinetic fatigue protocol followed by assessments of passive and active joint position sense being more vulnerable. Understanding these changes will contribute to developing rehabilitation strategies focusing on proprioception and fatigue management.

We expect that isokinetic fatigue will impair proprioception, with active joint position

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 50-65
* Postmenopausal
* Grade 2-3 knee osteoarthritis (Kellgren-Lawrence Scale) for OA group
* No lower extremity surgery in the last 6 months
* No neuromuscular or orthopedic condition affecting the lower extremities

Exclusion Criteria:

* Severe balance disorders or vestibular disease
* Bilateral knee prosthesis or severe osteoporosis
* Lower extremity musculoskeletal injury in the last 6 months

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Joint Position Sense | From enrollment to the end of intervention for 10 minutes
  Passive Joint Position Sense Test:
  The knee joint will be passively moved to 45°, then returned to the starting position. The participant will be asked to perceive and replicate the same angle passively. The difference between the perceived and actual angles will be recorded. An isokinetic dynamometer will be used during this test.
  Active Joint Position Sense Test:
  With their eyes closed, participants will be asked to actively move their knee to 45° and then return to the starting position. They will then be asked to actively reproduce the same angle. The difference between the measured and target angles will be recorded. An isokinetic dynamometer will be used during this test.

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.